CLINICAL TRIAL: NCT02543918
Title: Vaccination Response Following Administration of Ixekizumab to Healthy Subjects
Brief Title: A Study of the Immune Response to Vaccines and Ixekizumab (LY2439821) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16202; I1F-MC-RHCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
MeSH Terms: interventions — ixekizumab; Boostrix; Tetanus Toxoid; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ixekizumab + Boostrix® + Pneumovax®23 (Experimental): Ixekizumab administered once by subcutaneous injection (SQ) at week 0 and once at week 2.
  Boostrix® and Pneumovax®23 administered once by intramuscular (IM) injection into opposing arms at week 2.
  Interventions: Drug: Ixekizumab; Drug: Boostrix®; Drug: Pneumovax®23
- Boostrix® + Pneumovax®23 (Other): Boostrix® and Pneumovax®23 administered once by IM injection into opposing arms at week 2.
  Interventions: Drug: Boostrix®; Drug: Pneumovax®23

INTERVENTIONS:
Drug: Ixekizumab — Administered by SQ injection
  Other Names: LY2439821
  Arms: Ixekizumab + Boostrix® + Pneumovax®23
Drug: Boostrix® — Administered by IM injection
  Other Names: Tetanus, diphtheria, acellular pertussis vaccine (Tdap)
Drug: Pneumovax®23 — Administered by IM injection
  Other Names: Pneumococcal polysaccharide vaccine

SUMMARY:
The purpose of this study is to compare the body's immune response when vaccines are given alone versus when vaccines are given along with the study drug called ixekizumab. The vaccines protect against pneumonia and tetanus. This study will last about 6 weeks with follow-up at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females without compromised immune system
* Have a body mass Index of 18 to 32 kilograms per square meter (kg/m²)

Exclusion Criteria:

* Previously completed or withdrawn from an ixekizumab study or a study investigating interleukin-17 (IL-17) antagonists
* Have participated, within the last 30 days, in a clinical trial involving an investigational product. If the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed
* Have known allergy or hypersensitivity to any biologic therapy
* Past vaccination allergy or Arthus-type hypersensitivity
* Received a tetanus toxoid-containing vaccine within the last 5 years
* Severe allergic reaction to Boostrix
* Allergic to latex
* Have been immunized with pneumococcal vaccine
* Known hypogammaglobulinemia
* History of Guillain-Barre Syndrome
* Active infectious disease
* Had a live vaccination within 1 year prior to screening, or intend to have a live vaccination during the course of the study
* Evidence of a significant uncontrolled neuropsychiatric disorder -
* Have a score of 3 on Item 12 of the Quick Inventory of Depressive Symptomatology-Self Report (16 Items) at screening
* Evidence of Human Immunodeficiency Virus infection, Hepatitis C, B
* Had symptomatic herpes zoster within 3 months of screening
* Women who are lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Covance, Daytona Beach, Florida
  - Covance, Evansville, Indiana
  - Covance, Dallas, Texas

REFERENCES:
- [Derived] Gomez EV, Bishop JL, Jackson K, Muram TM, Phillips D. Response to Tetanus and Pneumococcal Vaccination Following Administration of Ixekizumab in Healthy Participants. BioDrugs. 2017 Dec;31(6):545-554. doi: 10.1007/s40259-017-0249-y. PMID 29116597

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixekizumab + Boostrix® + Pneumovax®23: Ixekizumab administered once by subcutaneous injection (SQ) at week 0 and once at week 2.
  Boostrix® and Pneumovax®23 administered once by IM injection into opposing arms at week 2.
- Boostrix® + Pneumovax®23: Boostrix® and Pneumovax®23 administered once by intramuscular (IM) injection into opposing arms at week 2.
Period: Overall Study
Arm/Group | Ixekizumab + Boostrix® + Pneumovax®23 | Boostrix® + Pneumovax®23
Started | 41 | 43
Received at Least 1 Dose of Study Drug | 41 | 42
Completed | 38 | 39
Not Completed | 3 | 4
Not completed — Never treated | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ixekizumab + Boostrix® + Pneumovax®23: Ixekizumab administered once by SQ at week 0 and once at week 2. Boostrix® and Pneumovax®23 administered once by IM injection into opposing arms at week 2.
- Total: Total of all reporting groups
Arm/Group | Ixekizumab + Boostrix® + Pneumovax®23 | Boostrix® + Pneumovax®23 | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (12.2) | 39.5 (10.5) | 41.4 (11.5)
Gender [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 22 | 24 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 34 | 35 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 17 | 32
  White | 24 | 25 | 49
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 84

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Immune Response to Tetanus and Pneumococcal Vaccinations
Description: Responder to tetanus vaccine defined as a post-vaccination anti-tetanus antibody concentration of >=1.0 (International Unit (IU) and a >=1.5-fold increase (50% increase) from baseline if the pre-vaccination concentration is <=1.0 at baseline OR a >=2.5-fold increase (150% increase) from baseline if the pre-vaccination concentration is > 1.0 IU at baseline.
  Responder to the pneumococcal vaccine is defined as a >=2-fold increase (100% increase) from baseline in anti-pneumococcal antibody concentrations against >50% of the 23 serotypes.
Time Frame: Week 6
Population: All randomized participants who completed the study.
Measure: Number; unit: percentage of participants
Arm/Group | Ixekizumab + Boostrix® + Pneumovax®23 | Boostrix® + Pneumovax®23
Number analyzed (Participants) | 38 | 41
percentage of participants
  Tetanus Vaccine Responders | 52.6 | 51.2
  Pneumococcal Vaccine Responders | 89.5 | 90.2
Statistical Analysis 1: Comparison: Ixekizumab + Boostrix® + Pneumovax®23 vs Boostrix® + Pneumovax®23; Tetanus vaccine responders; Test type: Non-Inferiority or Equivalence — Noninferiority of the ixekizumab arm to the control arm for the tetanus vaccine was established if the lower limit of the 90% CI excludes an absolute difference of 40% or more; Mean Difference (Final Values) = 1.4, 90% CI 2-sided [-16.6 to 19.2]
Statistical Analysis 2: Comparison: Ixekizumab + Boostrix® + Pneumovax®23 vs Boostrix® + Pneumovax®23; Pneumococcal vaccine responders; Test type: Non-Inferiority or Equivalence — Noninferiority of the ixekizumab arm to the control arm for the pneumococcal vaccine was established if the lower limit of the 90% CI excludes an absolute difference of 40% or more; Mean Difference (Final Values) = -0.8, 90% CI 2-sided [-12.9 to 11.0]

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | Ixekizumab + Boostrix® + Pneumovax®23 | Boostrix® + Pneumovax®23
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 1/41 | 0/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ixekizumab + Boostrix® + Pneumovax®23 (N=41) | Boostrix® + Pneumovax®23 (N=42)
Vulvovaginal candidiasis (Infections and infestations) | 1/19 (1) | 0/18 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less